CLINICAL TRIAL: NCT00789178
Title: Cognitive and Memory Function in Patients With Fibromyalgia and Their Influence on Disability
Brief Title: Cognitive and Memory Function in Patients With Fibromyalgia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Prof. Moshe Tishler /Head Department of Medicine B, Asaf Harofe Medical Center
Other Study IDs: 154/08
Record Dates: First submitted 2008-11-09; First posted 2008-11-11 (Estimated); Last update posted 2008-11-11 (Estimated); Status verified 2008-11

CONDITIONS: Fibromyalgia; Cognitive Impairment
Keywords: memory disturbances
MeSH Terms: conditions — Fibromyalgia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with fibromyalgia
- patients with active RA

SUMMARY:
Patients suffering from Fibromyalgia will be examined for the presence of memory and/or cognitive impairment using specific psychological tests.

Their results will be compared to those with active RA associated with pain and with a normal control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from fibromyalgia patients suffering from active RA

Exclusion Criteria:

* Patients with depressive disorders Patients treated with SSRI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 patients with fibromyalgia 30 patients with RA 20 healthy controls
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-10 (Estimated); Study Completion 2010-04 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Asaf Harofe Medical Center, Zrifin, Israel